CLINICAL TRIAL: NCT00409370
Title: A Randomized Clinical Trial to Compare The Use Of Safety Net Enclosures With Standard Restraints in Agitated Hospitalized Patients
Brief Title: Trial of Safety Nets In Hospitalized Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Griffin Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2002-25
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2006-12-08 (Estimated); Status verified 2006-12

CONDITIONS: Delirium; Agitated Behavior; Alcohol Withdrawl; Acute Confusional State; Acute Psychosis
MeSH Terms: conditions — Delirium; Psychomotor Agitation

INTERVENTIONS:
Device: SOMA safe enclosure

SUMMARY:
This study compared standard hospital restraints to a newer safety net restraint system to compare them for acceptability, tolerance, duration of restrain, length of stay in the hospital, and satisfaction of MD, nurse, and relatives of patients.

ELIGIBILITY:
Inclusion Criteria:

1. age more than 18
2. hospitalized
3. acute confusion or agitation

Exclusion Criteria:

1. Patients who require acute respiratory or cardiac support such as patients requiring ventilator support or patients in cardiac or septic shock
2. Patients who have a documented history of claustrophobia
3. Patients or family members who refuse to consent for safety net treatment under any circumstances. Failure to obtain consent due to absence of or inability to reach a family member or to give consent to participate in the study
4. Failure to obtain consent due to absence of or inability to reach a family member within reasonable time or to give consent to participate in the study.
5. Acutely ill patients requiring intravenous vasopressors, intubation or ventilatory support
6. Other conditions deemed terminal within 24 hours as determined by the patient's attending physician
7. Patients who stay less than 24 hours in the hospital
8. If patient is already on restrains for more than 48 hours preceding enrollment.
9. If two or more limbs are already on restraint to protect IV lines.
10. Extreme degree of agitation requiring continuous IV sedation or anesthesia. Such patients may pose a danger to staff or themselves if their restraints were to be discontinued in order to put them on study restraints.
11. When the intent of single wrist restraint is only to hold the IV line and patient is not agitated or in delirium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-04; Study Completion 2005-02

PRIMARY OUTCOMES:
Perception of the Nurse
perception of physician
perception of family member
agitated behavior scale
alcohol withdrawal assessment scale

SECONDARY OUTCOMES:
total duration of restraint use
length of hospital stay
total sedative medication dose used

CONTACTS AND LOCATIONS:
Overall Officials: haq nawaz, MD, Principal Investigator — Griffin Hospital
Locations (1):
- Griffin Hospital, Derby, Connecticut, United States